CLINICAL TRIAL: NCT07080320
Title: Research on the Evolution, Geometry, and Alterations of the Periorbital Region Based on Age and Deformations
Acronym: REGARD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2025_843_0101
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Facial Skin; Motion Capture; Aging; Periorbital Region; Skin Movement; Vertical Jump
Keywords: Facial skin; motion capture; aging; periorbital region; mechanical; skin movement; vertical jump

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subjects aged 18-33 years (Experimental)
  Interventions: Device: MoCap
- subjects aged 50-65 years (Experimental)
  Interventions: Device: MoCap

INTERVENTIONS:
Device: MoCap — For each subject, the displacement of markers, the deformation of regions between markers, and the evolution of angles formed by the markers during facial expressions and vertical movements will be analyzed with MoCap. These will be compared between the two age groups (18-33 years vs. 50-65 years) using a MANOVA model. The reference values for marker displacement will be defined by the interval between the 2.5% and 97.5% percentiles of the values for each marker. If the distribution is Gaussian, the percentiles will be derived from the standard normal distribution; otherwise, the non-parametric method will be used.
  The intervention will be Interventions :
  * Recruitment of healthy and pathological subjects.
  * Full-face and macro images of the periorbital region
  * Measurement of periorbital skin properties using MoCap and standard reference tools.
  * Application of a tightening product (aloe vera) and periorbital massage.
  * Measurement of skin response to a vertical jump.

SUMMARY:
The periorbital region of the face is a critical area affected by aging. Motion Capture (MoCap) allows the precise measurement of the mechanical properties of skin in this region. This study will validate MoCap as a tool for quantifying these properties, comparing it to traditional reference tools, and exploring how these properties evolve with age and external treatments. It will also assess MoCap's ability to detect the effects of various treatments such as tightening products and massages. Ultimately, this research will provide a deeper understanding of skin dynamics in the periorbital region and offer insights into both medical and cosmetic applications.

ELIGIBILITY:
Inclusion Criteria:

* Female participants
* Caucasian, Fitzpatrick skin types I-III
* BMI between 18.5 and 27, healthy participants
* Aged 18 to 65 years (inclusive)
* Not under guardianship or curatorship
* Informed written consent
* Social security affiliation
* Non-smokers for at least 5 years
* No excessive UV exposure (artificial or natural) in the last 3 weeks prior to the study or during the study

Exclusion Criteria:

* Severe skin disorders preventing the application of electrodes or photo-reflective markers
* Neurovascular history affecting the face
* Ongoing treatments influencing facial tissues (e.g., corticosteroids)
* Current sleep disorders
* Psychiatric conditions or social interaction impairments
* Inner ear or balance disorders
* Osteoporosis, recent fractures, or fragile bone conditions
* Pregnant or breastfeeding women
* Under guardianship, curatorship, or legal protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-09-20 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
maximum displacement (in millimeters) of each marker placed on the face | day 1
  maximum displacement (in millimeters) of each marker placed on the face during standardized movements of the periorbital region

SECONDARY OUTCOMES:
Coefficient of variation of the maximum displacement amplitudes measured during repeated tests for the same movement. | day 1
The correlation coefficient between dynamic MoCap measurements and static measurements obtained from reference tools. | day 1
  The correlation coefficient between dynamic MoCap measurements and static measurements obtained from reference tools.
The difference in the mean maximum displacement amplitudes (in millimeters) between different age groups | day 1
  The difference in the mean maximum displacement amplitudes (in millimeters) between different age groups
The difference in the mean maximum displacement amplitudes (in millimeters) before and after performing a periorbital massage | day 1
  The difference in the mean maximum displacement amplitudes (in millimeters) before and after performing a periorbital massage
The maximum mean displacement amplitudes (in millimeters) during a mechanical solicitation (a standardized vertical jump). | day 1
  The maximum mean displacement amplitudes (in millimeters) during a mechanical solicitation (a standardized vertical jump).
The difference in the mean maximum displacement amplitudes (in millimeters) before and after applying a tightening product (aloe vera). | day 1
  The difference in the mean maximum displacement amplitudes (in millimeters) before and after applying a tightening product (aloe vera).

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No